CLINICAL TRIAL: NCT05618288
Title: Impact of a Mobile Health Breastfeeding Counseling Intervention for Employed Mothers in Kenya
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wheaton College (Other)
Collaborators: Kenya Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ICKES221114
Record Dates: First submitted 2022-11-15; First posted 2022-11-16 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Breastfeeding, Exclusive
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Randomization to mobile health or in-person breastfeeding counseling
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): Standard of care breastfeeding counseling. The ongoing antenatal, delivery and postnatal breastfeeding and lactation counseling that is provided by the Naivasha sub-County Referral Hospital.
  Interventions: Behavioral: Standard of care breastfeeding counseling
- mobile Health (mHealth) (Experimental): Simple messaging service counseling intervention with healthcare providers. This arm will involve two-way messaging with healthcare providers Unstructured Supplementary Service Data application that provides session-based interaction with breastfeeding and lactation support content.
  Interventions: Behavioral: mobile Health Breastfeeding Counseling

INTERVENTIONS:
Behavioral: mobile Health Breastfeeding Counseling — a phone-based breastfeeding counseling intervention, delivered by labor and delivery nurses, nutritionists, and maternal and child health nurses.
  Arms: mobile Health (mHealth)
Behavioral: Standard of care breastfeeding counseling — The ongoing antenatal, delivery and postnatal breastfeeding and lactation counseling that is provided by the Naivasha sub-County Referral Hospital.
  Arms: Standard of Care

SUMMARY:
Exclusive breastfeeding (EBF) is critical for child survival, growth, and maternal health; however, over half of mothers in low and middle-income countries (LMIC). Mobile health (mHealth) describes a range of wireless technologies and techniques that seek to increase patient access to and interaction with preventive health services. This study will develop and test the feasibility of an mHealth intervention to improve support counseling for breastfeeding at a large sub-county referral hospital in Naivasha, Kenya.

DETAILED DESCRIPTION:
Exclusive breastfeeding (EBF) is critical for child survival, growth, and maternal health; however, over half of mothers in low and middle-income countries (LMICs) do not practice EBF through the recommended six months of infancy. Maternal employment is a significant risk factor for early cessation of EBF in LMICs. Policies in Kenya seek to support working mothers to continue practicing EBF after a nationally mandated 12-week maternity leave. However, the implementation of this policy is limited, and only 17% of formally employed mothers practice EBF through the recommended six months in Naivasha, Kenya, where a high proportion of mothers are employed in commercial agriculture and other low-wage industries.

Mobile health (mHealth) describes a range of wireless technologies and techniques that seek to increase patient access to and interaction with preventive health services. mHealth technologies hold untapped potential to support healthcare workers' training and counseling approaches to support lactation for working mothers, especially when collaboratively developed with end users.

This study will develop and test the feasibility of an mHealth intervention to improve support counseling for breastfeeding at a large sub-county referral hospital in Naivasha, Kenya. The primary objective of this proposal is to develop mHealth technology to equip and support healthcare worker breastfeeding counseling, and implement and evaluate its impact. We hypothesize that a culturally sensitive and technologically appropriate mHealth counseling intervention will improve EBF rates among infants of employed mothers. This study will be conducted in three aims:

Before the clinical trial phase of the study begins, we will employ a human-centered design approach to iteratively develop and test the feasibility of an mHealth intervention to support breastfeeding counseling for employed mothers.

After developing the technology, we will evaluate the impact of the mHealth breastfeeding counseling intervention on the outcomes of EBF, child morbidity, and worker presenteeism.

The overarching goal of this proposal is to develop an mHealth intervention that can successfully support continued lactation and BF for employed mothers across various sectors and be disseminated at a national scale in Kenya and other LMIC contexts where employed mothers face unique challenges to practicing EBF while maintaining employment.

Mothers will be recruited in the third trimester of pregnancy and followed through 9-months postpartum. 284 mothers will be randomly assigned to an mHealth counseling intervention or the Standard of Care (in person counseling at the Naivasha Sub-County Referral Hospital). there will be 142 mothers in each intervention arm.

ELIGIBILITY:
Inclusion Criteria:

* Mothers over 18 years who are employed in contract-based labor in sectors that include education, business, healthcare, commercial agriculture, tourism/food service.
* Mothers must reside in the greater Naivasha, Kenya area and receive maternal and child health care at the Naivasha sub-County Referral Hospital.

Exclusion Criteria:

* Mothers of infants with cleft deformities or other abnormalities that interfere with breastfeeding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 284 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2028-01-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Exclusive breastfeeding at 24 weeks | 24 weeks post-partum
  The proportion of mothers who feed only breastmilk to their infants, without other liquids, formula or semi-solid or solid food.

SECONDARY OUTCOMES:
Continued breastfeeding | 36 weeks post partum
  Any breastfeeding in the past 24 hours
Early initiation of breastfeeding | Within 1 hour of childbirth
  Breastfeeding within 1 hour of childbirth

CONTACTS AND LOCATIONS:
Overall Officials: Scott B Ickes, Principal Investigator — Wheaton College

IPD SHARING:
Plan to Share IPD: Yes
Only de-identified data will be shared with other researchers. This will include maternal research identification number, education level, martial status, parity, type of employment, child morbidity and breastfeeding status (at 0, 6, 14, 24, and 36 weeks weeks).
Supporting Information: Study Protocol, SAP
Time Frame: 2 months after the primary data analysis is complete.
Access Criteria: Permission of the principal investigator.